CLINICAL TRIAL: NCT00688610
Title: Antibiotics in Patients With Acute Respiratory Tract Infections in Primary Care in Consideration of Procalcitonin as Additive Parameter
Brief Title: Antibiotics in Patients With Acute Respiratory Tract Infection With Procalcitonin as Parameter
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Prof. Dr. med. Tobias Welte, Prof. Dr. med. Tobias Welte
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HannoverPro II
Record Dates: First submitted 2008-05-15; First posted 2008-06-03 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Respiratory Tract Infection
Keywords: primary care; procalcitonin; antibiotic prescription
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: laboratory value procalcitonin — A. attending physician includes patient with acute respiratory infection in study, indicates antibiotic prescription and collects procalcitonin-value. Waits for decision from laboratory either "change of decision" or "retention of decision". In case of "change decision": antibiotic is not recommended, patient shall not take antibiotic. In case of "retention of decision": patient may take the antibiotic.
  B. attending physician includes patient with acute respiratory infection in study, indicates NO antibiotic and collects procalcitonin-value. Waits for decision from laboratory either "change of decision" or "retention of decision". In case of "change decision": antibiotic is recommended, patient has to be informed about. In case of "retention of decision": no change.

SUMMARY:
Antibiotics in patients with acute respiratory tract infections in primary care in consideration of procalcitonin as additive parameter.

The purpose of this study is to compare the ordinary manner of antibiotic- prescription with the prescription in consideration of procalcitonin-value in patients with acute respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Informed consent
* Respiratory tract infection based on the clinical judgement of the primary care physician

Exclusion Criteria:

* Antibiotic pretreatment in previous 14 days
* Portal hypertension
* Major surgeries or multiple trauma which require hospitalization, in previous 4 weeks
* Autoimmune disease and systemic diseases (lupus erythematodes, wegener´s disease)
* Peritoneal dialysis
* Acute treated or recently operated medullary c-cell-carcinoma, SCLC, carcinoid
* Other inflammatory diseases (e.g. urinary tract infection, pyelonephritis, pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
days with significant impairment due to acute respiratory tract infection | 14 to 28 days after infection

SECONDARY OUTCOMES:
number of antibiotic prescriptions | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Burkhardt, Dr., Principal Investigator — Medical School Hannover
Locations (1):
- Medical School Hannover, Department Pneumology, Hanover, Germany

REFERENCES:
- [Derived] Burkhardt O, Ewig S, Haagen U, Giersdorf S, Hartmann O, Wegscheider K, Hummers-Pradier E, Welte T. Procalcitonin guidance and reduction of antibiotic use in acute respiratory tract infection. Eur Respir J. 2010 Sep;36(3):601-7. doi: 10.1183/09031936.00163309. Epub 2010 Feb 25. PMID 20185423